CLINICAL TRIAL: NCT01235962
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Pazopanib as Adjuvant Therapy for Subjects With Localized or Locally Advanced RCC Following Nephrectomy
Brief Title: A Study to Evaluate Pazopanib as an Adjuvant Treatment for Localized Renal Cell Carcinoma (RCC)
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113387; 2010-020965-26 (EudraCT Number); CPZP034D2301 (Other: Novartis)
Record Dates: First submitted 2010-10-14; First posted 2010-11-08 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Renal Cell Carcinoma (RCC); Cancer
Keywords: anti-angiogenic agent; renal cell carcinoma; pazopanib; adjuvant therapy; VEGFR inhibitor; localized or locally; advanced renal cell carcinoma (RCC) following nephrectomy; advanced RCC; Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pazopanib (Experimental): Pazopanib oral agent, administered at 600 mg daily initial dose for 8-12 weeks. Dose can be escalated to 800 mg daily based on safety evaluation. Complete treatment is 12 months. Dose can be reduced, interrupted or discontinued due to adverse events or intolerance.
  Interventions: Drug: pazopanib
- placebo (Placebo Comparator): placebo matching pazopanib 200 mg tablets, administered at 600 mg daily initial dose for 8-12 weeks. Dose can be escalated to 800 mg daily based on safety evaluation. Complete treatment is 12 months. Dose can be reduced, interrupted or discontinued due to adverse events or intolerance.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pazopanib — Pazopanib monohydrochloride salt was supplied as aqueous, film-coated tablets containing 200 mg of the free base. The 200 mg tablets were oval-shaped and white in color.
  Other Names: PZP034
  Arms: pazopanib
Drug: placebo — Placebo matching pazopanib was supplied as aqueous, film-coated tablets containing 200 mg of the free base. The 200 mg tablets were oval-shaped and white in color.
  Arms: placebo
Drug: pazopanib — Pazopanib 600 mg daily initial dose for 8-12 weeks, dose can be escalated to 800 mg daily based on safety evaluation.
  Other Names: Votrient
  Arms: pazopanib
Drug: placebo — placebo matching pazopanib daily initial dose for 8-12 weeks, dose can be escalated to 800 mg daily based on safety evaluation.
  Arms: placebo

SUMMARY:
This randomized Phase III study is to evaluate whether pazopanib compared with placebo can prevent or delay recurrence of kidney cancer in patients with moderately high or high risk of developing recurrence after undergoing kidney cancer surgery.

DETAILED DESCRIPTION:
The primary objective of this ongoing study was to evaluate DFS with pazopanib 600 mg daily initial dose as compared with placebo as adjuvant therapy for subjects with localized/locally advanced RCC following nephrectomy.

Subjects with locally recurrent renal cell carcinoma (RCC), bilateral RCC, or history of another malignancy were excluded from enrolling in the study.

The study was comprised of three successive study periods: 1) the Screening/Baseline period, 2) the study treatment period, and 3) the DFS /OS follow-up period. The Screening/Baseline period had a maximum duration of 12 weeks from the date of nephrectomy to the date of randomization.

After a subject met all the eligibility criteria and completed all the required baseline assessments, the subject was randomized in a 1:1 ratio to receive once daily blinded treatment with either pazopanib 600 mg as initial dose or matching placebo based on pre-defined stratification factors.

Subjects received continuous daily treatment until completion of the 12-month treatment period, disease recurrence, or unacceptable toxicity/intolerance. Subsequent adjuvant therapies for RCC were not allowed. During the study treatment and DFS follow-up periods, subjects received routine safety and efficacy assessments.

The study treatment period was 12 months. Subjects received continuous daily treatment until completion of the 12 month treatment period, disease recurrence, or unacceptable toxicity/intolerance. Subsequent adjuvant therapies for RCC were not allowed.

All subjects, regardless of study treatment status (i.e. premature discontinuation or completion of the 12-month treatment), were to be followed with routine imaging assessments and remain blinded until objective evidence of disease recurrence was obtained or until the study achieved the required number of events for the primary endpoint of DFS (319 events). After objective evidence of disease recurrence was obtained, subjects could be unblinded and received the first-line treatment for metastatic RCC per local standard of care.

All subjects were off treatment for at least 4 years at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Diagnosis of RCC with clear-cell or predominant clear-cell histology
* Subjects with non-metastatic disease (M0) fulfilling any of the following combinations of pathologic staging based on American Joint Committee on Cancer (AJCC) TNM staging version 2010 and Fuhrman nuclear grading.

  * pT2, G3 or G4, N0; or,
  * pT3, G any, N0; or,
  * pT4, G any, N0; or,
  * pT any, G any, N1
* Fulfill all of the following criteria of disease-free status at baseline:

  * Had complete gross surgical resection of all RCC via radical or partial nephrectomy using either open or laparoscopic technique.
  * Baseline imaging of chest, abdomen and pelvis shows no metastasis or residual tumor lesions as confirmed centrally by an independent radiologist.
* Received no prior adjuvant or neo-adjuvant treatment for RCC
* Recovered from nephrectomy: any surgery related toxicities should be reduced to ≤ grade 1 per NCI Common Terminology Criteria for Adverse Events (CTCAE) (Version 4)
* Karnofsky performance scale (KPS) of ≥ 80
* Adequate organ system function

Exclusion Criteria:

* History of another malignancy. Exception: Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Active diarrhea of any grade
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* History of human immunodeficiency virus (HIV) infection
* History of active hepatitis
* Presence of uncontrolled infection.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
* History of Class III or IV congestive heart failure, as defined by the New York Heart Association Classification of Congestive Heart Failure
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Corrected QT interval (QTc) > 480 milliseconds (msec)
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study (see Section 7.6.2 for instruction on blood pressure measurement and obtaining mean blood pressure values).

* Evidence of active bleeding or bleeding diathesis
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study treatment and for the duration of the study.
* Concurrent therapy given to treat cancer including treatment with an investigational agent or concurrent participation in another clinical trial involving anti-cancer investigational drug.
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or excipients that in the opinion of the investigator contraindicates their participation.
* Prior or current use of systemic anti-VEGF inhibitors, cytokines (e.g. interferon, interleukin 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (257):
- United States (56):
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Antioch, California
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, South San Francisco, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Saint Louis Park, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Springfield, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Hampton, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Virginia Beach, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Argentina (10):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Aut6noma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Austria (4):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (6):
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Wilrijk
- Brazil (8):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Canada (12):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Chile (2):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, Región Metro de Santiago
- China (5):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (8):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava - Poruba
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Ústí nad Labem
- Denmark (3):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Dk-2730 Herlev
  - Novartis Investigative Site, Odense C
- France (16):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Germany (39):
  - Novartis Investigative Site, Kirchheim, Baden-Wurttemberg
  - Novartis Investigative Site, Ravensburg, Baden-Wurttemberg
  - Novartis Investigative Site, Sigmaringen, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Weiden, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Offenbach, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Bergisch Gladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Neuss, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Homburg, Saarland
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Plauen, Saxony
  - Novartis Investigative Site, Dessau, Saxony-Anhalt
  - Novartis Investigative Site, Eisleben Lutherstadt, Saxony-Anhalt
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Hamburg
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion, Crete
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szombathely
- Ireland (4):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, Tallaght, Dublin
- Israel (6):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Zrifin
- Italy (11):
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Rozzano (MI), Lombardy
  - Novartis Investigative Site, Candiolo (TO), Piedmont
  - Novartis Investigative Site, Arezzo, Tuscany
  - Novartis Investigative Site, Terni, Umbria
  - Novartis Investigative Site, Negrar, Veneto
- Japan (8):
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hokkaido
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Yamagata
- Novartis Investigative Site, Luxembourg, Luxembourg
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (13):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Žilina
- South Korea (6):
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Jeonju
  - Novartis Investigative Site, Seongnam-si Gyeonggi-do
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Songpa-gu, Seoul
- Spain (9):
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Dos Hermanas (Sevilla)
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Oviedo
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (8):
  - Novartis Investigative Site, Brighton
  - Novartis Investigative Site, Cornwall
  - Novartis Investigative Site, Guildford
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Swansea
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, Barrios CH, Salman P, Gladkov OA, Kavina A, Zarba JJ, Chen M, McCann L, Pandite L, Roychowdhury DF, Hawkins RE. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8. doi: 10.1200/JCO.2009.23.9764. Epub 2010 Jan 25. PMID 20100962
- [Derived] Motzer RJ, Russo P, Haas N, Doehn C, Donskov F, Gross-Goupil M, Varlamov S, Kopyltsov E, Lee JL, Lim HY, Melichar B, Zemanova M, Rini B, Choueiri TK, Wood L, Reaume MN, Stenzl A, Chowdhury S, McDermott R, Michael A, Izquierdo M, Aimone P, Zhang H, Sternberg CN; PROTECT study investigators. Adjuvant Pazopanib Versus Placebo After Nephrectomy in Patients With Localized or Locally Advanced Renal Cell Carcinoma: Final Overall Survival Analysis of the Phase 3 PROTECT Trial. Eur Urol. 2021 Mar;79(3):334-338. doi: 10.1016/j.eururo.2020.12.029. Epub 2021 Jan 15. PMID 33461782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to include 1500 subjects. A total of 1538 subjects were enrolled and analyzed.
Groups:
- ITT Pazopanib 800 mg: Pazopanib 800 mg daily dose based on safety evaluation. Complete treatment is 12 months.
- ITT Placebo 800 mg: Placebo matching pazopanib 800 mg daily. Complete treatment is 12 months.
- ITT Pazopanib 600 mg: Pazopanib 600 mg daily initial dose for 8-12 weeks. Dose can be escalated to 800 mg daily based on safety evaluation. Complete treatment is 12 months.
- ITT Placebo 600 mg: Placebo matching pazopanib 600 mg daily. Complete treatment is 12 months.
Period: Overall Study
Arm/Group | ITT Pazopanib 800 mg | ITT Placebo 800 mg | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Started | 198 | 205 | 571 | 564
Prem. Withdrawn = Did Not Complete Study | 46 | 35 | 118 | 86
All Deaths | 43 | 46 | 102 | 104
Completed (Completed means dead or completed survival follow-up until the study completed.) | 152 | 170 | 453 | 478
Not Completed | 46 | 35 | 118 | 86
Not completed — Withdrawal by Subject | 20 | 19 | 62 | 49
Not completed — Lost to Follow-up | 21 | 16 | 47 | 32
Not completed — Physician Decision | 5 | 0 | 9 | 5

BASELINE CHARACTERISTICS:
Population: ITT 800 included all randomized subjects with a scheduled initial dose of 800 mg daily.
  ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
  Total (ITT All) included all randomized subjects, i.e. subjects either with a scheduled initial dose of 600 or 800 mg daily.
Groups:
- Total: Total of all reporting groups
Arm/Group | ITT Pazopanib 800 mg | ITT Placebo 800 mg | ITT Pazopanib 600 mg | ITT Placebo 600 mg | Total
Number analyzed (Participants) | 198 | 205 | 571 | 564 | 1538
Age, Customized [Number; unit: Participants]
  =>18 to <65 | 154 | 140 | 430 | 406 | 1130
  =>65 to <75 | 36 | 55 | 122 | 131 | 344
  =>75 to <85 | 8 | 10 | 19 | 27 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 51 | 173 | 164 | 447
  Male | 139 | 154 | 398 | 400 | 1091
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 168 | 178 | 471 | 481 | 1298
  Asian | 28 | 26 | 71 | 70 | 195
  African American/African Heritage | 1 | 0 | 7 | 1 | 9
  Other | 0 | 1 | 4 | 2 | 7
  Missing | 1 | 0 | 18 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) With Pazopanib 600 mg Daily Initial Dose vs. Placebo
Description: DFS is defined as the interval between the date of randomization and the earliest date of disease recurrence/metastasis or death due to any cause.
Time Frame: approximately 5 years
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
months | NA [NA to NA] — NA = DFS median and confidence interval were not determined because not enough events occurred at the analysis | NA [NA to NA] — NA = DFS median and confidence interval were not determined because not enough events occurred at the analysis
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.1649, Stratified Log-Rank; Adjusted Hazard Ratio = 0.862, 95% CI 2-sided [0.699 to 1.063]

2. Secondary Outcome: Overall Survival (OS) With Pazopanib 600 mg Daily Initial Dose vs. Placebo
Description: Overall survival is defined as the time from randomization until death due to any cause.
  For subjects who did not die, time to death was censored at the last date of known contact.
Time Frame: approximately 8.5 years
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
months | 89.5 [NA to NA] — NA = the last follow-up patient in this group died at the end of study, so the median survival was estimated (the survival curve crossed 50%). But the 95% CI was not estimable due to less than 50% events (death) occurring in pazopanib group. | NA [NA to NA] — NA = the last follow-up patient in this group was censored at the end of study and less than 50% events (death) occurred, so both median and 95%CI were not estimable
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.9880, Stratified Log-Rank; Adjusted Hazard Ratio = 0.998, 95% CI 2-sided [0.759 to 1.311]

3. Secondary Outcome: DFS Rates at Yearly Time Points With Pazopanib 600 mg Daily Initial Dose vs. Placebo
Time Frame: yearly for 4 years
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
Proportion of participants
  DFS at 1 year: number analyzed (Participants) | 423 | 394
  DFS at 1 year | 0.85 [0.81 to 0.88] | 0.76 [0.72 to 0.79]
  DFS at 2 years: number analyzed (Participants) | 308 | 300
  DFS at 2 years | 0.72 [0.67 to 0.75] | 0.68 [0.64 to 0.72]
  DFS at 3 years: number analyzed (Participants) | 118 | 118
  DFS at 3 years | 0.65 [0.61 to 0.70] | 0.64 [0.59 to 0.68]
  DFS at 4 years: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: DFS With Pazopanib vs. Placebo
Description: as for outcome 1
Time Frame: approximately 5 years
Population: Total (ITT All) included all randomized subjects, i.e. subjects either with a scheduled initial dose of 600 or 800 mg daily.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ITT All - Pazopanib: All randomized subjects with a scheduled initial dose of 600 or 800 mg daily pazopanib.
- ITT All - Placebo: All randomized subjects with a scheduled initial dose of 600 or 800 mg daily placebo.
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
months | NA [NA to NA] — NA = DFS median or confidence interval were not determined because not enough events occurred at the analysis. | NA [48.1 to NA] — NA = DFS median or upper limit of confidence interval were not determined because not enough events occurred at the analysis.
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.0126, Stratified Log-Rank; Adjusted Hazard Ratio = 0.802, 95% CI 2-sided [0.675 to 0.954]

5. Secondary Outcome: OS With Pazopanib vs. Placebo
Description: Overall survival is defined as the time from randomization until death due to any cause.
  For subjects who do not die, time to death will be censored at the last date of known contact.
Time Frame: approximately 8.5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
months | NA [NA to NA] — NA = OS median or confidence interval were not determined because not enough events occurred at the analysis. | NA [NA to NA] — NA = OS median or confidence interval were not determined because not enough events occurred at the analysis.
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.9959, Stratified Log-Rank; Adjusted Hazard Ratio = 1.001, 95% CI 2-sided [0.796 to 1.257]

6. Secondary Outcome: DFS Rates at Yearly Time Points With Pazopanib vs. Placebo
Time Frame: yearly for 4 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
Proportion of participants
  DFS at 1 year: number analyzed (Participants) | 579 | 538
  DFS at 1 year | 0.85 [0.82 to 0.87] | 0.75 [0.72 to 0.78]
  DFS at 2 years: number analyzed (Participants) | 436 | 419
  DFS at 2 years | 0.72 [0.68 to 0.75] | 0.66 [0.63 to 0.70]
  DFS at 3 years: number analyzed (Participants) | 231 | 215
  DFS at 3 years | 0.65 [0.62 to 0.69] | 0.61 [0.58 to 0.65]
  DFS at 4 years: number analyzed (Participants) | 48 | 46
  DFS at 4 years | 0.62 [0.58 to 0.66] | 0.56 [0.51 to 0.61]

7. Secondary Outcome: DFS Pazopanib 800 mg Daily Initial Dose vs. Placebo
Description: as for outcome 1
Time Frame: approximately 5 years
Population: ITT 800 included all randomized subjects with a scheduled initial dose of 800 mg daily.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITT Pazopanib 800 mg | ITT Placebo 800 mg
Number analyzed (Participants) | 198 | 205
months | NA [NA to NA] — NA = DFS median or confidence interval were not determined because not enough events occurred at the analysis. | 48.1 [30.1 to NA] — NA = DFS median or upper limit confidence interval were not determined because not enough events occurred at the analysis.
Statistical Analysis 1: Comparison: ITT Pazopanib 800 mg vs ITT Placebo 800 mg; Test type: Superiority; p = 0.0201, Stratified Log-Rank; Adjusted Hazard Ratio = 0.693, 95% CI 2-sided [0.510 to 0.943]

8. Secondary Outcome: OS With Pazopanib 800 mg Daily Initial Dose vs. Placebo
Description: as for outcome 2
Time Frame: approximately 8.5 years
Population: ITT 800 included all randomized subjects with a scheduled initial dose of 800 mg daily.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITT Pazopanib 800 mg | ITT Placebo 800 mg
Number analyzed (Participants) | 198 | 205
months | NA [NA to NA] — NA = OS was not determined because not enough events occurred at the analysis. | NA [NA to NA] — NA = OS was not determined because not enough events occurred at the analysis.
Statistical Analysis 1: Comparison: ITT Pazopanib 800 mg vs ITT Placebo 800 mg; Test type: Superiority; p = 0.9865, Stratified Log-Rank; Adjusted Hazard Ratio = 1.004, 95% CI 2-sided [0.662 to 1.521]

9. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using NCCN/Functional Assessment of Cancer Therapy-Kidney Symptom Index -19 (FACT FKSI-19) Total Score
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains (FKSI-DRS-P, FKSI-DRS-E, FKSI-TSE, FKSI-FWB) experienced in the past 7 days. Participants are asked to respond to a total of 19 questions regarding symptoms, side effects, and well being by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total score of 0 to 76). A negative mean indicates a worsening of condition. DFS: disease-free survival; FU: follow up
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52: number analyzed (Participants) | 423 | 401
  Week 52 | -3.83 (0.452) | -0.43 (0.459)
  24M DFS FU: number analyzed (Participants) | 335 | 340
  24M DFS FU | 0.19 (0.419) | 0.23 (0.418)
  36M DFS FU: number analyzed (Participants) | 294 | 290
  36M DFS FU | -0.14 (0.454) | -0.26 (0.456)
  48M DFS FU: number analyzed (Participants) | 144 | 140
  48M DFS FU | -0.13 (0.526) | 0.22 (0.529)
  54M DFS FU: number analyzed (Participants) | 60 | 66
  54M DFS FU | 0.09 (0.653) | 0.26 (0.635)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -3.397, 95% CI 2-sided [-4.486 to -2.307]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.930, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU) = -0.043, 95% CI 2-sided [-1.003 to 0.917]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.828, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.119, 95% CI 2-sided [-0.958 to 1.196]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.603, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = -0.347, 95% CI 2-sided [-1.658 to 0.964]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.841, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = -0.170, 95% CI 2-sided [-1.843 to 1.503]

10. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using NCCN/FACT FKSI-19 Scale Disease-related Symptoms-physical (DRS-P) Domain Score
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The DRS-P domain assesses symptoms experienced in the past 7 days. Participants are asked to respond to 12 questions ("I have a lack of energy," "I feel pain," for example) by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 48). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52: number analyzed (Participants) | 427 | 406
  Week 52 | -2.06 (0.278) | -0.44 (0.282)
  24M DFS FU: number analyzed (Participants) | 340 | 341
  24M DFS FU | -0.32 (0.273) | -0.20 (0.273)
  36M DFS FU: number analyzed (Participants) | 300 | 293
  36M DFS FU | -0.61 (0.291) | -0.53 (0.294)
  48M DFS FU: number analyzed (Participants) | 147 | 141
  48M DFS FU | -0.67 (0.332) | -0.46 (0.336)
  54M DFS FU: number analyzed (Participants) | 61 | 66
  54M DFS FU | -0.21 (0.449) | -0.55 (0.439)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -1.619, 95% CI 2-sided [-2.283 to -0.955]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.726, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24 M DFS FU) = -0.114, 95% CI 2-sided [-0.750 to 0.522]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.801, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36 M DFS FU) = -0.090, 95% CI 2-sided [-0.789 to 0.609]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.617, analysis of covariance; adjusted for baseline score using mixed-model; Meat Difference (48 M DFS FU) = -0.212, 95% CI 2-sided [-1.044 to 0.320]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.565, adjusted for baseline score using mixedm; Mean Difference (54 M DFS FU) = 0.341, 95% CI 2-sided [-0.828 to 1.510]

11. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using NCCN/FACT FKSI-19 Scale Disease Related Symptoms-emotional (DRS-E) Domain Score
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The DRS-E domain assesses symptoms experienced in the past 7 days. Participants are asked to respond to the question of "I worry that my condition will get worse" by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 4). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU,48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52: number analyzed (Participants) | 425 | 402
  Week 52 | 0.01 (0.054) | 0.09 (0.055)
  24M DFS FU: number analyzed (Participants) | 338 | 340
  24M DFS FU | 0.11 (0.056) | 0.16 (0.056)
  36M DFS FU: number analyzed (Participants) | 296 | 291
  36M DFS FU | 0.13 (0.059) | 0.12 (0.059)
  48M DFS FU: number analyzed (Participants) | 146 | 141
  48M DFS FU | 0.08 (0.075) | 0.20 (0.076)
  54M DFS FU: number analyzed (Participants) | 60 | 66
  54M DFS FU | 0.04 (0.090) | 0.24 (0.087)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.238, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -0.077, 95% CI 2-sided [-0.205 to 0.051]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.442, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU) = -0.052, 95% CI 2-sided [-0.185 to 0.081]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.819, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.016, 95% CI 2-sided [-0.125 to 0.158]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.223, analysis of covariance; analysis of covariance adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = -0.119, 95% CI 2-sided [-0.311 to 0.073]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.085, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = -0.203, 95% CI 2-sided [-0.435 to 0.028]

12. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using NCCN/FACT FKSI-19 Scale Treatment Side Effects (TSE) Domain Score
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The TSE domain assesses side effects experienced in the past 7 days. Participants are asked to respond to 3 questions ("I have nausea," "I have diarrhea," and "I am bothered by side effects of treatment") by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 12). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU,48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52: number analyzed (Participants) | 426 | 404
  Week 52 | -1.73 (0.101) | -0.34 (0.103)
  24M DFS FU: number analyzed (Participants) | 338 | 341
  24M DFS FU | 0.12 (0.061) | 0.01 (0.060)
  36M DFS FU: number analyzed (Participants) | 299 | 292
  36M DFS FU | 0.05 (0.067) | -00.3 (0.067)
  48M DFS FU: number analyzed (Participants) | 146 | 140
  48M DFS FU | -0.04 (0.087) | -0.01 (0.088)
  54M DFS FU: number analyzed (Participants) | 61 | 66
  54M DFS FU | 0.07 (0.089) | 0.09 (0.086)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -1.394, 95% CI 2-sided [-1.660 to -1.129]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.083, analysis of covariance; adjusted for baseline score using mixed-model; Mean difference (24M DFS FU) = 0.117, 95% CI 2-sided [-0.015 to 0.249]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.307, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.081, 95% CI 2-sided [-0.074 to 0.236]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.796, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = -0.029, 95% CI 2-sided [-0.249 to 0.191]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.885, analysis of covariance; adjusted for baseline score using mixed-models; Mean Difference (54M DFS FU) = -0.016, 95% CI 2-sided [-0.237 to 0.205]

13. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using NCCN/FACT FKSI-19 Scale Functional Well Being (FWB) Domain Score
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The FWB domain assesses well being in the past 7 days. Participants are asked to respond to 3 questions ("I am able to work," "I am able to enjoy life," and "I am content with the quality of my life now") by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 12). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU,48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52: number analyzed (Participants) | 426 | 406
  Week 52 | 0.06 (0.153) | 0.33 (0.155)
  24M DFS FU: number analyzed (Participants) | 339 | 341
  24M DFS FU | 0.39 (0.168) | 0.32 (0.168)
  36M DFS FU: number analyzed (Participants) | 299 | 293
  36M DFS FU | 0.43 (0.177) | 0.24 (0.178)
  48M DFS FU: number analyzed (Participants) | 146 | 141
  48M DFS FU | 0.51 (0.219) | 0.42 (0.222)
  54M DFS FU: number analyzed (Participants) | 61 | 66
  54M DFS FU | 0.31 (0.308) | 0.59 (0.299)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.143, analysis of covariance; adjusted for baseline score using mixed-model; Mean Differencec (Week 52) = -0.270, 95% CI 2-sided [-0.633 to 0.092]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.736, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU) = 0.069, 95% CI 2-sided [-0.336 to 0.475]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.397, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.188, 95% CI 2-sided [-0.247 to 0.623]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.781, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = 0.081, 95% CI 2-sided [-0.488 to 0.649]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.503, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = -0.278, 95% CI 2-sided [-1.094 to 0.539]

14. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib 600 mg Daily Initial Dose vs. Placebo Assessed Using EuroQoL-5D (EQ-5D) Score
Description: Health outcome and quality of life measured by EQ-5D thermometer (thermo) score and EQ-5D utility index (UI) score. The EQ-5D is a participant-answered questionnaire measuring 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D has two separate components: utility score and thermometer score. The EQ-5D total utility score ranges from 0 (worst health state) to 1 (perfect health state); 1 reflects the best outcome. The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: ITT 600 included all randomized subjects with a scheduled initial dose of 600 mg daily.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT Pazopanib 600 mg | ITT Placebo 600 mg
Number analyzed (Participants) | 571 | 564
scores on a scale
  Week 52 thermo. score: number analyzed (Participants) | 417 | 399
  Week 52 thermo. score | 0.713 (0.858) | 1.430 (0.868)
  24M DFS FU thermo. score: number analyzed (Participants) | 328 | 334
  24M DFS FU thermo. score | 3.356 (0.882) | 3.641 (0.877)
  36M DFS FU thermo. score: number analyzed (Participants) | 288 | 287
  36M DFS FU thermo. score | 3.640 (0.882) | 2.459 (0.883)
  48M DFS FU thermo. score: number analyzed (Participants) | 144 | 141
  48M DFS FU thermo. score | 3.909 (1.014) | 3.184 (1.015)
  54M DFS FU thermo. score: number analyzed (Participants) | 60 | 65
  54M DFS FU thermo. score | 3.076 (1.607) | 1.053 (1.560)
  Week 52 UI score: number analyzed (Participants) | 419 | 401
  Week 52 UI score | -0.019 (0.009) | -0.001 (0.009)
  24M DFS FU UI score: number analyzed (Participants) | 334 | 337
  24M DFS FU UI score | -0.004 (0.010) | 0.016 (0.010)
  36M DFS FU UI score: number analyzed (Participants) | 294 | 288
  36M DFS FU UI score | 0.002 (0.011) | -0.008 (0.011)
  48M DFS FU UI score: number analyzed (Participants) | 144 | 141
  48M DFS FU UI score | -0.002 (0.013) | 0.008 (0.013)
  54M DFS FU UI score: number analyzed (Participants) | 61 | 65
  54M DFS FU UI score | 0.004 (0.017) | -0.013 (0.017)
Statistical Analysis 1: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.490, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52 thermo) = -0.717, 95% CI 2-sided [-2.751 to 1.318]
Statistical Analysis 2: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.788, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU- thermo) = -0.285, 95% CI 2-sided [-2.358 to 1.788]
Statistical Analysis 3: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.266, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU- thermo) = 1.180, 95% CI 2-sided [-0.901 to 3.262]
Statistical Analysis 4: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.570, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU - thermo) = 0.725, 95% CI 2-sided [-1.779 to 3.229]
Statistical Analysis 5: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.346, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU - thermo) = 2.023, 95% CI 2-sided [-2.205 to 6.251]
Statistical Analysis 6: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.111, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52 - UI) = -0.018, 95% CI 2-sided [-0.040 to 0.004]
Statistical Analysis 7: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.094, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU - UI) = -0.020, 95% CI 2-sided [-0.044 to 0.003]
Statistical Analysis 8: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.490, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU - UI) = 0.010, 95% CI 2-sided [-0.018 to 0.037]
Statistical Analysis 9: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.580, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU - UI) = -0.009, 95% CI 2-sided [-0.043 to 0.024]
Statistical Analysis 10: Comparison: ITT Pazopanib 600 mg vs ITT Placebo 600 mg; Test type: Superiority; p = 0.473, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU - UI) = 0.017, 95% CI 2-sided [-0.029 to 0.063]

15. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using National Comprehensive Cancer Network (NCCN)/FACT FKSI-19 Total Score
Description: as for outcome 9
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52: number analyzed (Participants) | 575 | 554
  Week 52 | -4.01 (0.385) | -0.47 (0.388)
  24M DFS FU: number analyzed (Participants) | 462 | 458
  24M DFS FU | 0.23 (0.361) | 0.33 (0.362)
  36M DFS FU: number analyzed (Participants) | 405 | 392
  36M DFS FU | 0.16 (0.385) | -0.07 (0.389)
  48M DFS FU: number analyzed (Participants) | 244 | 232
  48M DFS FU | 0.47 (0.421) | 0.39 (0.427)
  54M DFS FU: number analyzed (Participants) | 156 | 153
  54M DFS FU | 0.27 (0.505) | -0.14 (0.509)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -3.536, 95% CI 2-sided [-4.466 to -2.606]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.812, analysis of covariance; adjusted for baseline score using mixed-model; Mean difference (24M DFS FU) = -0.102, 95% CI 2-sided [-0.942 to 0.738]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.621, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.233, 95% CI 2-sided [-0.690 to 1.155]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.878, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = 0.082, 95% CI 2-sided [-0.959 to 1.122]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.533, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = 0.412, 95% CI 2-sided [-0.887 to 1.712]

16. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using National Comprehensive Cancer Network (NCCN)/FACT FKSI-19 Scale Disease-related Symptoms-physical (DRS-P) Domain Score
Description: Health outcome and quality of life measured by NCCN/FACT FKSI-19 questionnaire for ITT ALL. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The DRS-P domain assesses symptoms experienced in the past 7 days. Participants are asked to respond to 12 questions ("I have a lack of energy," "I feel pain," for example) by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 48). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52: number analyzed (Participants) | 579 | 559
  Week 52 | -2.03 (0.235) | -0.51 (0.237)
  24M DFS FU: number analyzed (Participants) | 467 | 460
  24M DFS FU | -0.24 (0.232) | -0.25 (0.233)
  36M DFS FU: number analyzed (Participants) | 412 | 395
  36M DFS FU | -0.41 (0.247) | -0.45 (0.250)
  48M DFS FU: number analyzed (Participants) | 248 | 233
  48M DFS FU | -0.25 (0.270) | -0.19 (0.275)
  54M DFS FU: number analyzed (Participants) | 157 | 153
  54M DFS FU | -0.23 (0.329) | -0.68 (0.333)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -1.515, 95% CI 2-sided [-2.078 to -0.952]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.961, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU) = 0.014, 95% CI 2-sided [-0.534 to 0.561]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.888, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.043, 95% CI 2-sided [-0.555 to 0.641]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.858, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = -0.061, 95% CI 2-sided [-0.736 to 0.614]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.300, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = 0.452, 95% CI 2-sided [-0.404 to 1.309]

17. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using National Comprehensive Cancer Network (NCCN)/FACT FKSI-19 Scale Disease-related Symptoms-emotional (DRS-E) Domain Score
Description: Health outcome and quality of life measured by NCCN/FACT FKSI-19 questionnaire for ITT ALL. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The DRS-E domain assesses symptoms experienced in the past 7 days. Participants are asked to respond to the question of "I worry that my condition will get worse" by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 4).A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52: number analyzed (Participants) | 578 | 555
  Week 52 | 0.04 (0.045) | 0.14 (0.046)
  24M DFS FU: number analyzed (Participants) | 465 | 458
  24M DFS FU | 0.15 (0.048) | 0.19 (0.048)
  36M DFS FU: number analyzed (Participants) | 407 | 393
  36M DFS FU | 0.19 (0.050) | 0.15 (0.051)
  48M DFS FU: number analyzed (Participants) | 246 | 243
  48M DFS FU | 0.16 (0.059) | 0.20 (0.060)
  54M DFS FU: number analyzed (Participants) | 156 | 153
  54M DFS FU | 0.16 (0.065) | 0.17 (0.066)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.059, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52) = -0.103, 95% CI 2-sided [-0.211 to 0.004]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.487, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU) = -0.041, 95% CI 2-sided [-0.155 to 0.074]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.885, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.037, 95% CI 2-sided [-0.085 to 0.160]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.676, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = -0.032, 95% CI 2-sided [-0.183 to 0.119]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.859, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = -0.015, 95% CI 2-sided [-0.183 to 0.153]

18. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using National Comprehensive Cancer Network (NCCN)/FACT FKSI-19 Scale Treatment Side Effects (TSE) Domain Score
Description: Health outcome and quality of life measured by NCCN/FACT FKSI-19 questionnaire for ITT ALL. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The TSE domain assesses side effects experienced in the past 7 days. Participants are asked to respond to 3 questions ("I have nausea," "I have diarrhea," and "I am bothered by side effects of treatment") by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 12). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52: number analyzed (Participants) | 578 | 557
  Week 52 | -1.86 (0.089) | -0.33 (0.090)
  24M DFS FU: number analyzed (Participants) | 465 | 460
  24M DFS FU | 0.12 (0.052) | 0.04 (0.052)
  36M DFS FU: number analyzed (Participants) | 411 | 394
  36M DFS FU | 0.11 (0.057) | -0.02 (0.058)
  48M DFS FU: number analyzed (Participants) | 247 | 232
  48M DFS FU | 0.05 (0.065) | -0.00 (0.066)
  54M DFS FU: number analyzed (Participants) | 157 | 153
  54M DFS FU | 0.09 (0.074) | 0.03 (0.074)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p < .001, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (Week 52) = -1.535, 95% CI 2-sided [-1.769 to -1.300]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.127, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (24M DFS FU) = 0.089, 95% CI 2-sided [-0.025 to 0.202]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.069, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (36M DFS FU) = 0.123, 95% CI 2-sided [-0.009 to 0.255]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.544, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (48M DFS FU) = 0.049, 95% CI 2-sided [-0.110 to 0.208]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.518, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = 0.061, 95% CI 2-sided [-0.124 to 0.246]

19. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using National Comprehensive Cancer Network (NCCN)/FACT FKSI-19 Scale Functional Well Being (FWB) Domain Score
Description: Health outcome and quality of life measured by NCCN/FACT FKSI-19 questionnaire for ITT ALL. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains. The FWB domain assesses well being in the past 7 days. Participants are asked to respond to 3 questions ("I am able to work," "I am able to enjoy life," and "I am content with the quality of my life now") by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total domain score of 0 to 12). A negative mean indicates a worsening of condition.
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52: number analyzed (Participants) | 579 | 559
  Week 52 | -0.08 (0.134) | 0.30 (0.136)
  24M DFS FU: number analyzed (Participants) | 467 | 460
  24M DFS FU | 0.30 (0.147) | 0.41 (0.147)
  36M DFS FU: number analyzed (Participants) | 411 | 395
  36M DFS FU | 0.3 (0.151) | 0.29 (0.153)
  48M DFS FU: number analyzed (Participants) | 247 | 243
  48M DFS FU | 0.50 (0.179) | 0.38 (0.183)
  54M DFS FU: number analyzed (Participants) | 157 | 153
  54M DFS FU | 0.39 (0.206) | 0.44 (0.208)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.022, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (Week 52) = -0.374, 95% CI 2-sided [-0.695 to -0.053]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.567, analysis of covariance; adjusted for baseline score using mixed-model; Mean Diffeence (24M DFS FU) = -0.104, 95% CI 2-sided [-0.462 to 0.253]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.706, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU) = 0.072, 95% CI 2-sided [-0.302 to 0.446]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.612, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU) = 0.120, 95% CI 2-sided [-0.343 to 0.583]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.870, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU) = -0.045, 95% CI 2-sided [-0.587 to 0.496]

20. Secondary Outcome: Health-related Quality of Life (HRQoL) With Pazopanib vs. Placebo for ITT ALL Assessed Using EuroQoL-5D (EQ-5D) Score
Description: Health outcome and quality of life measured by using EQ-5D thermometer score and EQ-5D utility index (UI) score. The EQ-5D is a participant-answered questionnaire measuring 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D has two separate components: utility score and thermometer score. The EQ-5D total utility score ranges from 0 (worst health state) to 1 (perfect health state); 1 reflects the best outcome. The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Week 52, 24M DFS FU, 36M DFS FU, 48M DFS FU, 54M DFS FU
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ITT All - Pazopanib | ITT All - Placebo
Number analyzed (Participants) | 769 | 769
scores on a scale
  Week 52 thermo.: number analyzed (Participants) | 568 | 546
  Week 52 thermo. | 0.744 (0.733) | 2.859 (0.742)
  24M DFS FU thermo.: number analyzed (Participants) | 452 | 450
  24M DFS FU thermo. | 4.043 (0.741) | 4.296 (0.743)
  36M DFS FU thermo.: number analyzed (Participants) | 398 | 387
  36M DFS FU thermo. | 3.997 (0.774) | 3.150 (0.781)
  48M DFS FU thermo.: number analyzed (Participants) | 245 | 232
  48M DFS FU thermo. | 4.683 (0.863) | 4.552 (0.877)
  54M DFS FU thermos.: number analyzed (Participants) | 155 | 149
  54M DFS FU thermos. | 3.650 (1.028) | 3.249 (1.043)
  Week 52 UI score: number analyzed (Participants) | 571 | 548
  Week 52 UI score | -0.023 (0.008) | 0.003 (0.008)
  24M DFS FU UI score: number analyzed (Participants) | 460 | 453
  24M DFS FU UI score | 0.001 (0.008) | 0.017 (0.008)
  36M DFS FU UI score: number analyzed (Participants) | 404 | 387
  36M DFS FU UI score | 0.004 (0.009) | -0.004 (0.009)
  48M DFS FU UI score: number analyzed (Participants) | 244 | 231
  48M DFS FU UI score | -0.004 (0.010) | 0.010 (0.010)
  54M DFS FU UI score: number analyzed (Participants) | 156 | 147
  54M DFS FU UI score | -0.004 (0.012) | 0.003 (0.012)
Statistical Analysis 1: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.018, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52 - thermo.) = -2.116, 95% CI 2-sided [-3.872 to -0.359]
Statistical Analysis 2: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.778, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU - thermo) = -0.253, 95% CI 2-sided [-2.014 to 1.508]
Statistical Analysis 3: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.376, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU - thermo) = 0.847, 95% CI 2-sided [-1.030 to 2.724]
Statistical Analysis 4: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.905, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU - thermo) = 0.131, 95% CI 2-sided [-2.032 to 2.294]
Statistical Analysis 5: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.768, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU - thermo) = 0.401, 95% CI 2-sided [-2.269 to 3.071]
Statistical Analysis 6: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.007, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (Week 52 - UI) = -0.026, 95% CI 2-sided [-0.044 to -0.007]
Statistical Analysis 7: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.130, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (24M DFS FU - UI) = -0.016, 95% CI 2-sided [-0.036 to 0.005]
Statistical Analysis 8: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.520, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (36M DFS FU - UI) = 0.007, 95% CI 2-sided [-0.015 to 0.030]
Statistical Analysis 9: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.276, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (48M DFS FU - UI) = -0.014, 95% CI 2-sided [-0.040 to 0.011]
Statistical Analysis 10: Comparison: ITT All - Pazopanib vs ITT All - Placebo; Test type: Superiority; p = 0.665, analysis of covariance; adjusted for baseline score using mixed-model; Mean Difference (54M DFS FU - UI) = -0.007, 95% CI 2-sided [-0.037 to 0.024]

21. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of approx. 13 months (treatment duration ranged from 0 to to 13 months). Deaths post treatment survival follow up were collected after the on-treatment period, up to approx. 8.5 years. Participants who had not died after study drug discontinuation were censored: 82% of participants in the ITT 600 population and 78% of participants in the ITT 800 population.
Time Frame: approx. 13 months, approx. 8.5 years
Population: Safety 800: subjects who received at least one dose of study treatment in the ITT 800 population Safety 600: subjects who received at least one dose of study treatment in the ITT 600 population
Measure: Number; unit: participants
Groups:
- Safety Pazopanib 800 mg: Pazopanib 800 mg daily dose based on safety evaluation. Complete treatment is 12 months.
- Safety Placebo 800 mg: Placebo matching pazopanib 800 mg daily based on safety evaluation. Complete treatment is 12 months.
- Safety Pazopanib 600 mg: Pazopanib 600 mg daily dose based on safety evaluation. Complete treatment is 12 months.
- Safety Placebo 600 mg: Placebo matching pazopanib 600 mg daily based on safety evaluation. Complete treatment is 12 months.
Arm/Group | Safety Pazopanib 800 mg | Safety Placebo 800 mg | Safety Pazopanib 600 mg | Safety Placebo 600 mg
Number analyzed (Participants) | 198 | 204 | 568 | 558
participants
  Total Deaths | 43 | 46 | 102 | 104
  On-Treatment Deaths | 1 | 0 | 3 | 0
  Deaths post-treatment survival follow-up | 42 | 46 | 99 | 104

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 28 days after study drug discontinuation, for a maximum duration of approx. 13 months (treatment duration ranged from 0 to to 13 months).
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus up to 28 days post treatment.
Groups:
- I TT Pazopanib 600 mg: Pazopanib 600 mg daily initial dose for 8-12 weeks. Dose can be escalated to 800 mg daily based on safety evaluation. Complete treatment is 12 months.
Arm/Group | ITT Pazopanib 800 mg | ITT Placebo 800 mg | I TT Pazopanib 600 mg | ITT Placebo 600 mg | ITT All - Pazopanib | ITT All - Placebo
All-Cause Mortality (participants affected / at risk) | 1/198 | 0/204 | 3/568 | 0/558 | 4/766 | 0/762
Serious Adverse Events (participants affected / at risk) | 44/198 | 14/204 | 123/568 | 54/558 | 167/766 | 68/762
Other Adverse Events (participants affected / at risk) | 194/198 | 147/204 | 541/568 | 448/558 | 735/766 | 595/762
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ITT Pazopanib 800 mg (N=198) | ITT Placebo 800 mg (N=204) | I TT Pazopanib 600 mg (N=568) | ITT Placebo 600 mg (N=558) | ITT All - Pazopanib (N=766) | ITT All - Placebo (N=762)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0 | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1
Macular hole (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 2 | 0 | 2 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 3 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 4 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 2 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 3 | 1 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0 | 3 | 1 | 8 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Lung transplant rejection (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 3
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1
Superinfection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 15 | 0 | 51 | 2 | 66 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 12 | 0 | 13 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 3 | 0 | 3 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 4 | 0 | 4 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 3 | 0 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 2 | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 1 | 0 | 4 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 1 | 3 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ITT Pazopanib 800 mg (N=198) | ITT Placebo 800 mg (N=204) | I TT Pazopanib 600 mg (N=568) | ITT Placebo 600 mg (N=558) | ITT All - Pazopanib (N=766) | ITT All - Placebo (N=762)
Neutropenia (Blood and lymphatic system disorders) | 12 | 0 | 25 | 2 | 37 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 1 | 22 | 6 | 34 | 7
Hypothyroidism (Endocrine disorders) | 24 | 2 | 55 | 4 | 79 | 6
Abdominal pain (Gastrointestinal disorders) | 27 | 24 | 85 | 46 | 112 | 70
Abdominal pain upper (Gastrointestinal disorders) | 18 | 5 | 58 | 18 | 76 | 23
Constipation (Gastrointestinal disorders) | 17 | 17 | 28 | 38 | 45 | 55
Diarrhoea (Gastrointestinal disorders) | 129 | 48 | 361 | 139 | 490 | 187
Dyspepsia (Gastrointestinal disorders) | 17 | 13 | 43 | 17 | 60 | 30
Flatulence (Gastrointestinal disorders) | 8 | 6 | 32 | 18 | 40 | 24
Nausea (Gastrointestinal disorders) | 89 | 28 | 226 | 89 | 315 | 117
Stomatitis (Gastrointestinal disorders) | 23 | 10 | 55 | 23 | 78 | 33
Vomiting (Gastrointestinal disorders) | 37 | 8 | 95 | 21 | 132 | 29
Asthenia (General disorders) | 24 | 12 | 79 | 53 | 103 | 65
Fatigue (General disorders) | 74 | 53 | 222 | 144 | 296 | 197
Mucosal inflammation (General disorders) | 21 | 5 | 46 | 17 | 67 | 22
Oedema peripheral (General disorders) | 12 | 10 | 17 | 29 | 29 | 39
Pyrexia (General disorders) | 13 | 7 | 21 | 22 | 34 | 29
Nasopharyngitis (Infections and infestations) | 13 | 12 | 27 | 40 | 40 | 52
Upper respiratory tract infection (Infections and infestations) | 11 | 7 | 12 | 21 | 23 | 28
Alanine aminotransferase increased (Investigations) | 51 | 11 | 146 | 26 | 197 | 37
Aspartate aminotransferase increased (Investigations) | 48 | 5 | 129 | 22 | 177 | 27
Blood bilirubin increased (Investigations) | 8 | 5 | 32 | 6 | 40 | 11
Blood creatinine increased (Investigations) | 14 | 14 | 29 | 32 | 43 | 46
Platelet count decreased (Investigations) | 10 | 1 | 32 | 7 | 42 | 8
Weight decreased (Investigations) | 10 | 2 | 33 | 7 | 43 | 9
Decreased appetite (Metabolism and nutrition disorders) | 42 | 11 | 112 | 22 | 154 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 13 | 47 | 68 | 65 | 81
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 15 | 53 | 78 | 82 | 93
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 10 | 26 | 11 | 39 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 8 | 39 | 32 | 55 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 12 | 42 | 30 | 64 | 42
Dizziness (Nervous system disorders) | 26 | 17 | 50 | 52 | 76 | 69
Dysgeusia (Nervous system disorders) | 43 | 5 | 171 | 15 | 214 | 20
Headache (Nervous system disorders) | 58 | 35 | 139 | 78 | 197 | 113
Insomnia (Psychiatric disorders) | 10 | 8 | 29 | 28 | 39 | 36
Proteinuria (Renal and urinary disorders) | 14 | 5 | 24 | 2 | 38 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12 | 51 | 52 | 66 | 64
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 | 2 | 55 | 10 | 69 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 35 | 26 | 52 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 47 | 11 | 63 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 6 | 64 | 19 | 90 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 9 | 38 | 32 | 52 | 41
Hair colour changes (Skin and subcutaneous tissue disorders) | 90 | 9 | 232 | 28 | 322 | 37
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 42 | 8 | 103 | 24 | 145 | 32
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 17 | 25 | 41 | 37 | 58
Rash (Skin and subcutaneous tissue disorders) | 24 | 14 | 63 | 36 | 87 | 50
Hypertension (Vascular disorders) | 108 | 30 | 294 | 107 | 402 | 137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.